CLINICAL TRIAL: NCT01554410
Title: A Phase I Trial of Intensity Modulated Radiation Therapy With Concurrent Cisplatin and Escalating Gemcitabine for Locally Advanced Cervical Carcinoma
Brief Title: Intensity Modulated Radiation Therapy With Cisplatin and Gemcitabine to Treat Locally Advanced Cervical Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Loren Mell, MD, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD 100597
Record Dates: First submitted 2012-03-08; First posted 2012-03-15 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Cervical Carcinoma
Keywords: Cervical; Carcinoma; Gemcitabine; Gemzar; Cisplatin; IMRT; Radiation; External Beam; Brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Carcinoma | interventions — Radiotherapy, Intensity-Modulated; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMRT/Cisplatin/Gemcitabine (Experimental): All patients get IMRT with concurrent cisplatin & gemcitabine, with the dose of gemcitabine varying according to cohort
  Interventions: Radiation: Intensity Modulated Radiation Therapy (IMRT); Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Radiation: Intensity Modulated Radiation Therapy (IMRT) — 45 Gy in 25 daily fractions (1.8 Gy per fraction)
Drug: Cisplatin — Weekly infusion of 40 mg/m2 x 5 weeks (70 mg maximum)
Drug: Gemcitabine — Weekly infusion x 5 weeks at escalating dose levels (50mg/m2, 75mg/m2, 100mg/m2, and 125mg/m2)

SUMMARY:
The primary objective of the study is to identify the highest dose of gemcitabine that can be given safely with cisplatin and pelvic intensity modulated radiation therapy (IMRT) in women with locally advanced cervical cancer. The investigators hypothesis is that IMRT will reduce gastrointestinal and hematologic toxicity, permitting escalating doses of gemcitabine to be feasibly delivered in patients with locally advanced cervical cancer.

DETAILED DESCRIPTION:
Many studies have investigated multiagent chemotherapy as a means of intensifying treatment. The results of such trials indicate that gemcitabine has considerable activity against cervical cancer when given with cisplatin/RT, however, it is quite toxic. The predominant toxicities are gastrointestinal and hematologic. Methods to reduce gastrointestinal and hematologic toxicity during chemoradiotherapy could mitigate this toxicity and take advantage of the therapeutic benefits of gemcitabine

IMRT is an advanced radiation therapy delivery technique that reduces the amount of radiation given to normal tissues and may therefore reduce unwanted side effects. IMRT tries to lower the amount of radiation that normal tissues receive, while still delivering the desired amount of radiation to the cancer cells and other areas, such as lymph nodes. IMRT does this by using computers to design the best way to aim radiation at the tumor(s), while still delivering a radiation dose comparable to standard radiation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Histologically-proven, invasive primary carcinoma of the cervix.
* Disease Status: Stage IB2-IVA cervical cancer or stage I with biopsy-proven pelvic node metastases, positive surgical margins, or parametrial extension based upon standard diagnostic workup, including:
* History/physical examination
* Examination under anesthesia (if indicated)
* Biopsy
* Intravenous pyelogram and/or cystoscopy (if indicated)
* Colonoscopy, sigmoidoscopy, or rigid proctoscopy (if indicated)
* PA and lateral chest x-ray or chest CT
* CT or MRI of the pelvis
* PET, PET/CT, or PET/CT simulation (encouraged)
* Performance Level: Karnofsky Performance Status ≥ 60 - Peripheral ≥ ANC 1500/uL
* Platelet count ≥ 100,000/uL (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dL is acceptable)
* Serum creatinine ≤ 1.5 mg/dl
* Bilirubin (sum of conjugated + unconjugated) < 1.5 mg/dl, and
* SGPT (ALT) < 1.5 x upper limit of normal (ULN) for age, and
* SGOT (AST) < 1.5 x upper limit of normal (ULN) for age

Exclusion Criteria:

* Pregnancy or Breast-Feeding: Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events.(Note: Serum Pregnancy tests must be obtained in women of child bearing potential). Sexually active females may not participate unless they have agreed to use an effective contraceptive method (such as abstinence, diaphragm, condom, or intrauterine device) to prevent pregnancy for the duration of the study.
* Concomitant Medications, if taken within the last 28 days.
* Growth factor(s): Growth factors that support platelet or white cell number or function must not have been administered within the past 28 days.
* Erythropoietic drug(s): Erythropoietin or related hormones must not have been administered within the past 28 days.
* Infection: Patients who have an uncontrolled infection.
* Evidence of para-aortic lymphadenopathy or distant metastases
* Prior invasive malignancy (except non-melanomatous skin cancer), unless disease free for a minimum of 3 years.
* Prior systemic chemotherapy within the last three years.
* Prior radiotherapy to the pelvis
* Allergic to iodinated contrast if undergoing a contrast enhanced CT scan of the pelvis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-08; Primary Completion 2019-07-16 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose (MTD) of Gemcitabine that can be safely administered in combination with Cisplatin | 5 weeks during treatment
  To determine the maximum tolerated dose (MTD) of weekly gemcitabine that can be administered with concurrent weekly cisplatin and pelvic intensity modulated radiation therapy (IMRT) in women with locally advanced cervical cancer

SECONDARY OUTCOMES:
Number of Participants with Acute Adverse Events as a Measure of Safety and Tolerability | Up to 30 Days post-treatment
  To quantify acute treatment-related adverse events that occur within 30 days of completing protocol treatment.
Number of Participants with Progression-Free Survival as a Measure of Response | Up to 12 months post treatment
  To determine the progression-free and overall survival of patients treated with gemcitabine at the MTD in this regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Loren Mell, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Moores UC San Diego Cancer Center, La Jolla, California, United States

REFERENCES:
- [Derived] Mell LK, Xu R, Yashar CM, McHale MT, Einck JP, Mayadev J, Lee E, Binder P, Rash D, Eskander R, Heide ES, Plaxe SC, Mundt AJ, Saenz CC. Phase 1 Trial of Concurrent Gemcitabine and Cisplatin with Image Guided Intensity Modulated Radiation Therapy for Locoregionally Advanced Cervical Carcinoma. Int J Radiat Oncol Biol Phys. 2020 Aug 1;107(5):964-973. doi: 10.1016/j.ijrobp.2020.04.019. Epub 2020 Apr 22. PMID 32334034